CLINICAL TRIAL: NCT04806919
Title: Randomized Controlled Trial Comparing Micronized Progesterone (Amelgen ®) 400 mg BID Versus 400 mg TID for Luteal Support in Artificial Vitrified/Warmed Single Blastocyst Transfer Cycles With Low Progesterone on Day of Embryo Transfer
Brief Title: Luteal Support in Artificial Vitrified/Warmed Cycles With Low Progesterone
Acronym: PROTECTA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-004112-10
Record Dates: First submitted 2021-01-18; First posted 2021-03-19 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: IVF; Embryo Loss; Luteal Phase Defect
MeSH Terms: conditions — Embryo Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Amelgen ® 400 mg BID (No Intervention): Continue daily dose progesteron
- Intervention group: Amelgen ® 400 mg TID (Experimental): Increase daily progesteron dose
  Interventions: Drug: Progesteron TID

INTERVENTIONS:
Drug: Progesteron TID — increasing the dose
  Arms: Intervention group: Amelgen ® 400 mg TID

SUMMARY:
The study aims to evaluate the effect of an increased dose of vaginal progesterone supplementation on the incidence of ongoing pregnancy for patients with a suboptimal serum progesterone level (defined as < 10 mcg/l) on the day of blastocyst transfer.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent form (ICF) dated and signed
* Age ≥ 18 and < 43 years old
* Body Mass Index (BMI) ≥ 18.5 kg/m2 and < 35 kg/m2
* Less than 4 previous Assisted Reproductive Technologies (ART) cycles
* Current pregnancy wish
* Patients undergoing a single vitrified/warmed single transfer in an artificial prepared endometrium cycle (IVF or ICSI)

Exclusion Criteria:

* Simultaneous participation in another clinical study
* Previous participation in this study
* Known reasons for impaired implantation (specifically: presence of a hydrosalpinx; presence of a type I, II or III fibroid; Asherman's syndrome; uterine malformations, intrauterine adhesions, ≥ grade 3 endometriosis according to the ASRM classification, endometrial tuberculosis)
* Repeated miscarriages (> 2 miscarriages)
* Untreated and uncontrolled thyroid dysfunction
* Tumors of the ovary, breast, uterus, pituitary or hypothalamus
* Abnormal vaginal bleeding without a known/diagnosed cause
* Ovarian cysts or enlarged ovaries
* Fibroid tumors of the uterus incompatible with pregnancy
* Malformations of the reproductive organs incompatible with pregnancy
* Previous antibiotic hypersensitivity reactions (streptomycin and/or neomycin)
* Risk factors for thromboembolic events, such as a personal or family history, severe obesity or thrombophilia
* Active smoking
* Ongoing pregnancy
* Use of carbamazepine, rifampicin or phenytoin
* Those unable to comprehend the investigational nature of the proposed study

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 242 (Estimated)
Dates: Start 2021-04-02 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 7 gestational weeks (+ or - 1 week)
  visualization of an embryo with a heart beat

SECONDARY OUTCOMES:
Endometrial impaction: Corelation between the change in endometrial thickness on day of embryo transfer and ongoing pregnancy rate | 7 gestational weeks (+ or - 1 week)

OTHER OUTCOMES:
Questionnaire on patient comfort and side effects | On the day of embryo transfer (day 5)
Questionnaire on patient comfort and side effects | On the day of the initial pregnancy test (day 16 (± 2 days))

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - UZ Ghent, Ghent
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No